CLINICAL TRIAL: NCT03670797
Title: Prevalence Of Oral Mucosal Alterations In a Sample of Egyptian Patients With Diabetes Mellitus Type2: A Hospital Based Cross Sectional Study
Brief Title: Prevalence Of Oral Mucosal Alterations In Diabetes Mellitus Type2
Status: Completed | Type: Observational
Sponsor: Alaa Mahmoud abd El kader (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Alaa Mahmoud abd El kader, principle investigator, internal resident at oral medicine department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Diabetes-Oral Alterations
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Oral Disease; Diabetes
Keywords: oral health status; oral findings; oral manifestations; patients with diabetes
MeSH Terms: conditions — Mouth Diseases; Diabetes Mellitus; Oral Manifestations

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- controlled diabetic patients
- uncontrolled diabetic patients

SUMMARY:
There are severe deficiency of database concerning the oral health status in Egyptian patients with Diabetes type 2. Our aim in the present study is to study the prevalence of oral mucosal alterations in type 2 DM patients and the effect of hyperglycemia on these alterations in controlled and uncontrolled patients to increase their awareness and minimize all the possible risk factors,to achieve a proper management for all oral problems.

DETAILED DESCRIPTION:
The study will be held in the Endocrine clinic at El Kasr Al-Ainy Cairo University Hospital for patients with diabetes mellitus type2. The data collected through the questionnaire will be obtained through an interview between the investigator and the patient.Clinical examination will be performed for the oral cavity.Blood sample will be withdrawn from each participant and collected in the clinical pathology lab in El kasr Al Ainy to measure the glycosylated hemoglobin concentration.The salivary gland function will be determined through a small questionnaire and clinical examination of the patient.

Selection bias: will be minimized by enrolling the participants in the study in a consecutive order of the entering the clinic.

Non-respondent bias: will be minimized by explaining to the participants the aim of the study and their importance and role in the study.

Incomplete records: will be excluded from statistical analysis with reporting the cause of not completing the record.

Sample size estimation:

Based on the previous papers by AL-Maweri,et al ,2013, the prevalence of oral mucosal alterations in diabetic patients 45.1%.Using a precision of 5, a design effect set at 1 with 95% CI (confidence interval), a total sample size of 381 will be sufficient. The sample size was calculated by Epi info.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Patients >25years old
3. Patients diagnosed with diabetes type 2.
4. Egyptian patients.

Exclusion Criteria:

1. females diagnosed with gestational diabetes.
2. Patients not physically able to participate in survey or clinical oral examination.
3. Patients with other systemic diseases which may cause oral manifestation as liver disorders.
4. Patients under immunosuppressive drugs.
5. Patients under corticosteriods.
6. Patients with organ transplantation.

Ages: 25 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A convenience sample of adult patients diagnosed with diabetes type 2 attending at the Endocrine clinic at El Kasr Al-Ainy Cairo University Hospital will be enrolled in the study in a consecutive order.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Oral mucosal alterations | 10 min
  Clinical examination according to WHO guidelines by Dichotomous outcome (Yes/No).

SECONDARY OUTCOMES:
Periodontal condition | 10 min
  Basic periodontal examination by Continuous outcome (Score codes).
Salivary glands function | 10 min
  Clinical oral dryness examination and Self estimated questionnaire by Dichotomous outcome (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Mariam fakhr, Study Chair — the Endocrine units at the Kasr Al-Ainy Cairo university hospital.
Locations (1):
- Alaa Mahmoud Abd El Kader, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Al-Maweri SA, Ismail NM, Ismail AR, Al-Ghashm A. Prevalence of oral mucosal lesions in patients with type 2 diabetes attending hospital universiti sains malaysia. Malays J Med Sci. 2013 Jul;20(4):39-46. PMID 24043995
- [Result] Bastos AS, Leite AR, Spin-Neto R, Nassar PO, Massucato EM, Orrico SR. Diabetes mellitus and oral mucosa alterations: prevalence and risk factors. Diabetes Res Clin Pract. 2011 Apr;92(1):100-5. doi: 10.1016/j.diabres.2011.01.011. Epub 2011 Mar 3. PMID 21300417